CLINICAL TRIAL: NCT02778087
Title: Self-directed Box (Mirror) Therapy After Stroke: A Dosing Study
Brief Title: Mirror Therapy After Stroke: A Dosing Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Helen Hayes Hospital (Other)
Responsible Party: Principal Investigator, Glen Gillen, Associate Professor of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAQ2004
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Stroke
Keywords: motor recovery; mirror therapy; upper extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAU plus 30 minutes of BT. (Experimental): Intervention: Subjects randomized to the 30 minute intervention will perform the above 15 minute Mirror Box Therapy intervention independently two times per day in addition to their treatment as usual.
  Interventions: Behavioral: Mirror Box Therapy
- TAU plus 60 minute of BT. (Experimental): Intervention: Subjects randomized to the 60 minute intervention will perform the above 15 minute Mirror Box Therapy intervention independently four times per day in addition to their treatment as usual.
  Interventions: Behavioral: Mirror Box Therapy
- TAU plus 30 minutes of sham BT. (Sham Comparator): Intervention: Subjects randomized to the control (sham) group will perform the above Sham Mirror Box Therapy intervention independently two times per day. The control group will be using a mirror box with an opaque surface as opposed to a reflective mirror.
  Interventions: Behavioral: Sham Mirror Box Therapy

INTERVENTIONS:
Behavioral: Mirror Box Therapy — The BT intervention will be delivered in 15 minute increments via a self-directed program. The subject will sit comfortably at a table or desk in front of a box, which will be positioned in the mid-sagittal plane. The subject will place his or her affected arm inside the box so that it is out of view. The subject will then place his or her unaffected arm on the table and will be instructed to focus their attention on the mirror reflection of the unaffected arm throughout the intervention. The 15 minute intervention will consist of the following movements/tasks: active range of motion (AROM), functional tasks with objects, and object manipulation.
  Arms: TAU plus 30 minutes of BT.; TAU plus 60 minute of BT.
Behavioral: Sham Mirror Box Therapy — The BT intervention will be delivered in 15 minute increments via a self-directed program. The subject will sit comfortably at a table or desk in front of a box, which will be positioned in the mid-sagittal plane. The subject will place his or her affected arm inside the box so that it is out of view. The subject will then place his or her unaffected arm on the table and will be instructed to focus their attention on an opaque mirror throughout the intervention. The 15 minute intervention will consist of the following movements/tasks: AROM, functional tasks with objects, and object manipulation.
  Arms: TAU plus 30 minutes of sham BT.

SUMMARY:
It has been suggested that augmenting repetitive task practice with the use of box (mirror) therapy (BT) can enhance the benefits of task practice and may provide stroke survivors an opportunity to engage in self-directed practice outside of normally scheduled therapy sessions. However, the dosage of BT to be used in clinical practice is unclear. In order for practitioners to begin integrating BT into clinical practice situations more information is needed to determine what defines a therapeutic dose. The aim of this study is to differentiate between two dosages of self-directed BT added to treatment as usual for decreasing arm and hand motor impairments, improving activity level, and increasing self-directed participation after stroke. Forty-five subjects from the Stroke Rehabilitation Unit at Helen Hayes Hospital (HHH) will be randomly assigned into three groups: treatment as usual plus 30 minute dosage of self-directed BT 5x/week; treatment as usual plus 60 minute dosage of self-directed BT 5x/week; treatment as usual plus 30 minutes of self-directed sham BT 5x/week.

DETAILED DESCRIPTION:
Approximately 795,000 people in the United States have a stroke each year, and stroke is considered a leading cause of long-term disability. Impairments in arm and hand function are common after stroke and limit engagement in daily life activities, which impacts the overall quality of life of stroke survivors. It has been found that incomplete upper limb recovery predicted health related quality of life in stroke survivors at one year post-stroke in four (self-care, usual activities, pain/discomfort, & anxiety/depression) out of five domains measured on the EuroQol-5D questionnaire. Thus, evidence-based interventions that improve arm and hand function after stroke are needed. In fact, a recent study identified "treatments for upper extremity recovery" to be one of the top ten research priorities relating to life after stroke according to stroke survivors, caregivers, and health professionals. Evidence suggests task-oriented training interventions such as Repetitive Task Practice (RTP) are effective at improving upper extremity (UE) function and activity, and therapy participation in stroke survivors.

Recently, it has been suggested that augmenting RTP with the use of cognitive strategies, such as Mirror Box Therapy (BT), can enhance the benefits of task practice and may provide stroke survivors an opportunity to engage in self-directed practice outside of normally scheduled therapy sessions. During BT, a person engages in motor activities with the unimpaired limb while watching its mirror reflection superimposed over the (unseen) impaired limb; this process creates a visual illusion whereby activities performed by the unimpaired limb are attributed to the impaired limb. While generating this visual illusion is a common ingredient in published BT effectiveness trials, the actual treatment protocols differ considerably. One important protocol difference seen across published trials relates to the dosage of BT. For instance, the minutes of BT provided range from 10 minutes to 60 minutes per session; session frequencies range from 1 to 7 sessions per week, and the length of the intervention ranges from 3 to 6 weeks. Thus, the dosage of BT to be used in clinical practice is unclear. In order for practitioners to begin integrating BT into clinical practice more information is needed on the effective dosage, as this may vary according to multiple factors (e.g., stage of recovery, the survivor's current functional limitations, or environment in which services are rendered).

ELIGIBILITY:
Inclusion Criteria:

* Adults status post ischemic or hemorrhagic stroke between the ages 18-85, receiving inpatient rehabilitation
* Using the impaired arm, ability to lift and release a wash cloth off a table with any means of prehension in either the sitting or standing positions
* A score > 21/30 on the Mini-Mental State Exam
* Ability to consent.

Exclusion Criteria:

* Serious visual or visual-perceptual deficits, neuropsychological impairments, or orthopedic conditions that would prevent participation in the BT protocol as determined by the treatment team
* Involvement in another study protocol related to motor function after stroke
* Anticipated length of stay less than two weeks
* More than six months post stroke

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01; Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Score on Action Research Arm Test: | pre and post intervention up to 12 months
  This test examines hand and arm motor function. It consists of 19 movement tasks divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale, ranging from 3 (performs test normally) to 0 (can perform no part of test). Totaled scores range from 0-57 with higher scores indicating higher functioning. Normative data for stroke has been published for this tool (Beebe & Lang, 2009; van der Lee et al., 2001). This tool has been found to be a valid measure (Platz et al., 2005; van der Lee et al., 2001). This test has excellent test-retest reliability (Platz et al., 2005), as well as inter-rater reliability (Nijland et al., 2010). Minimally clinically important difference (MCID) for this test has been established for both acute (Lang et al., 2008) and chronic stroke survivors (van der Lee et al., 2001).

SECONDARY OUTCOMES:
Score on Stroke Impact Scale | pre and post intervention up to 12 months
  This is a questionnaire including questions regarding whether the stroke has resulted in physical problems, problems with memory and thinking, changes in mood and emotions, problems with communication, daily living skills, mobility, and hand function. Normative data has been published for stroke survivors (Duncan et al., 2002). Several authors have established the validity of this tool (Doyle et al., 2007; Duncan et al., 2002; Huang et al., 2010; Kwon et al., 2006). This measure has adequate to excellent test-retest reliability depending on the domain (Duncan et al., 1999), as well as intra-rater reliability (Carod-Artal et al., 2009).
Score on Functional Independence Measure | pre and post intervention up to 12 months
  This provides a measurement of a subject's disability based on the International Classification of Impairment, Disabilities and Handicaps, and it indicates how much assistance the individual will need to carry out common basic activities of daily living. It contains 18 items that are rated on a seven point ordinal scale from total assistance to complete independence, and totaled scores range from a low of 18 to a high of 126, with higher scores indicating higher functioning. Normative data has been published for stroke survivors (Inouye et al., 2001). The validity of this measure has established (Inouye et al., 2001; Denti et al., 2008; Hsueh et al., 2002). This test has been found to have excellent test-retest reliability (Pollak et al., 1996; Hobart et al., 2001).
Score on Fugl-Meyer Assessment of Motor Recovery after Stroke (arm/hand section) | pre and post intervention up to 12 months
  This test examines a variety of reaching patterns, wrist and hand function, quality of movement, sensation, and reflexes. Items are scored on a 3-point ordinal scale from 0 (cannot perform) to 2 (performs fully). The domains assessed include: Motor function (UE maximum score = 66), Sensory function (UE maximum score = 12), and Joint pain (maximum score = 24). This tool is one of the most widely used quantitative measures of motor impairment after stroke (Gladstone et al., 2002). Multiple authors have documented the validity of this tool (Malouin et al., 1994; Mao et al., 2002; Shelton et al., 2001). It has excellent inter- and intra-rater reliability (Duncan, 1983). It has been found to be a strong predictor of motor function (Duncan, et al., 1992).

CONTACTS AND LOCATIONS:
Overall Officials: Glen Gillen, EdD, OTR, Principal Investigator — Columbia University; Steven W. Lichtman, EdD, Study Director — Helen Hayes Hospital
Locations (1):
- Helen Hayes Hospital (Stroke Unit), West Haverstraw, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsen DM, Gillen G, Geller D, Hreha K, Osei E, Saleem GT. Effectiveness of interventions to improve occupational performance of people with motor impairments after stroke: an evidence-based review. Am J Occup Ther. 2015 Jan-Feb;69(1):6901180030p1-9. doi: 10.5014/ajot.2015.011965. PMID 25553742
- [Background] Nilsen DM, DiRusso T. Using mirror therapy in the home environment: a case report. Am J Occup Ther. 2014 May-Jun;68(3):e84-9. doi: 10.5014/ajot.2014.010389. PMID 24797202
- [Background] Thieme H, Mehrholz J, Pohl M, Behrens J, Dohle C. Mirror therapy for improving motor function after stroke. Stroke. 2013 Jan;44(1):e1-2. doi: 10.1161/strokeaha.112.673087. PMID 23390640
- [Background] Thieme H, Mehrholz J, Pohl M, Behrens J, Dohle C. Mirror therapy for improving motor function after stroke. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD008449. doi: 10.1002/14651858.CD008449.pub2. PMID 22419334
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374